CLINICAL TRIAL: NCT03024242
Title: Tight Vaginoscopy: a Simplified Novel Technique for a Better Vaginal Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Khairy Ali, Lecturer, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: TVS
Record Dates: First submitted 2017-01-15; First posted 2017-01-18 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Endosalpingiosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tight vaginoscope (Experimental): The vaginoscope was extracted and loaded inside a thick rubber ring before its reinsertion inside the vagina again. To avoid leakage from the center of the thick rubber ring, the vaginoscopy is inserted through a premade central cruciate incision.
  Interventions: Device: Tight vaginoscope

INTERVENTIONS:
Device: Tight vaginoscope

SUMMARY:
Bivalve vaginal speculum insertion is a basic final step of vaginal examination. Unfortunately, it can't be inserted in young girls, virgins, nulliparous women with narrow vagina, women with vaginismus or patients with a history of previous vaginal surgery. In such cases, the value of vaginoscopy (examination of the vagina without speculum) is evident. Indications of vaginoscopy are expanding. In addition to confirmation of suspected vaginal masses or polypi diagnosis, it can be used to diagnose laceration of the vaginal wall in girls due to foreign body , traumatic injuries or sexual abuse. In a systematic review, the effectiveness and feasibility of using hysteroscopy for exploration of the immature genital tract (vaginoscopy) were documented.It may help in the diagnosis and treatment of gynecologic disorders in adolescent patients with an intact hymen, limited vaginal access, or a narrow vagina. Another recent systematic review highlighted the importance of Vagino-hysteroscopy as an easy way to gain access to the cervical canal and an important tool with which to diagnose and treat vaginal lesions.

In practice, we notice leakage of excessive irrigating fluid per vagina with poor visualization during vaginoscopy. To the best of our knowledge, no study addressed a solution to improve visualization and success of vaginoscopic surgery. This study aims to test feasibility and doctor satisfaction of performing conventional diagnostic vaginoscopy if compared to tight diagnostic vaginoscopy and success on performing tight vaginoscopic surgery in patients with vaginal or cervical lesions.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatizing women with suspected narrow vagina.
* Nulliparous women or virgin w
* Vaginal or cervical lesion or foreign body.

Exclusion Criteria:

* Multiparous women
* Nulliparous women with patulous or lax vaginae were excluded.

Ages: 10 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2014-07; Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
The success rate of the procedure | 20 minutes

SECONDARY OUTCOMES:
The satisfaction rate by satisfaction score | 20 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Women Health Hospital - Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes